CLINICAL TRIAL: NCT03493256
Title: Novel BIochemical Markers for Predicting Type 2 NEurological Complications of Surgical Coronary Revascularization (BINER): a Prospective Cohort Study.
Brief Title: Novel BIochemical Markers for Predicting Type 2 NEurological Complications of Surgical Coronary Revascularization (BINER)
Acronym: BINER
Status: Completed | Type: Observational
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Krzysztof Szwed, Principal Investigator, Collegium Medicum w Bydgoszczy
Other Study IDs: KB 776/2017
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Neurological Complication of Procedure (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type 2 neurological complications present: The group of patients diagnosed with postoperative cognitive dysfunction (POCD) or postoperative delirium (POD), or both concurrently.
  Interventions: Other: exposure to type 2 neurological complications
- type 2 neurological complications absent: The group of patients without neurological complications.

INTERVENTIONS:
Other: exposure to type 2 neurological complications — exposure to postoperative cognitive dysfunction (POCD) or postoperative delirium (POD), or both concurrently.
  Groups: type 2 neurological complications present

SUMMARY:
In this single center prospective cohort study a total of 100 patients scheduled for elective off-pump CABG will be recruited. They will be allocated to one study and one control group according to the presence or absence of postoperative type 2 neurological complications. The two groups will be compared in terms of serum concentrations of glial fibrillary acidic protein (GFAP), neuroserpin (NSP), phosphorylated axonal neurofilament subunit H (pNfH) and visinin-like protein 1 (VILIP-1) at the time of skin incision and closure as well as 24 hours and 7 days following surgery. Diagnostic performance of these markers for predicting type 2 neurological complications of off-pump CABG will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective off-pump Coronary Artery Bypass Grafting (CABG)

Exclusion Criteria:

* neurological or psychiatric disorders
* alcohol or drug abuse
* preoperative left ventricular ejection fraction of less than 30%
* extracranial carotid artery stenosis of more than 70%
* scoring below age- and education-adjusted cut-off values in Mini-Mental State Examination (MMSE)
* scoring over seven points on the subscales of the Hospital Anxiety and Depression Scale (HADS)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All participants will be recruited from patients scheduled for elective off-pump CABG at the Department of Cardiac Surgery, Dr Antoni Jurasz Memorial University Hospital, Bydgoszcz, Poland.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of serum GFAP concentration (ng/ml) changes. | GFAP concentrations will be measured preoperatively (at the time of initial skin incision), at the completion of surgery (at the time of skin closure) as well as 24 hours and 7 days following off-pump Coronary Artery Bypass Grafting (CABG).
  Comparison of patients with and without type 2 neurological complications in respect to changes from baseline concentration of glial fibrillary acidic protein (GFAP).
Assessment of serum NSP concentration (ng/ml) changes. | NSP concentrations will be measured preoperatively (at the time of initial skin incision), at the completion of surgery (at the time of skin closure) as well as 24 hours and 7 days following off-pump Coronary Artery Bypass Grafting (CABG).
  Comparison of patients with and without type 2 neurological complications in respect to changes from baseline concentration of neuroserpin (NSP).
Assessment of serum pNfH concentration (ng/ml) changes. | pNfH concentrations will be measured preoperatively (at the time of initial skin incision), at the completion of surgery (at the time of skin closure) as well as 24 hours and 7 days following off-pump Coronary Artery Bypass Grafting (CABG).
  Comparison of patients with and without type 2 neurological complications in respect to changes from baseline concentration of neuroserpin phosphorylated axonal neurofilament subunit H (pNfH).
Assessment of serum VILIP-1 concentration (ng/ml) changes. | VILIP-1 concentrations will be measured preoperatively (at the time of initial skin incision), at the completion of surgery (at the time of skin closure) as well as 24 hours and 7 days following off-pump Coronary Artery Bypass Grafting (CABG).
  Comparison of patients with and without type 2 neurological complications in respect to changes from baseline concentration of visinin-like protein 1 (VILIP-1).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Szwed, Dr, Principal Investigator — Department of Clinical Neuropsychology, Nicolaus Copernicus University, Collegium Medicum.
Locations (1):
- Department of Cardiac Surgery, Dr Antoni Jurasz Memorial University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, CSR
Time Frame: Available without time limits.
Access Criteria: The data that support the findings of this study are available from the corresponding author upon reasonable request.